CLINICAL TRIAL: NCT07013162
Title: Efficacy of Diode Laser and Non-Surgical Periodontal Therapy in the Treatment of Periodontitis: A Clinical and Immunological Study
Brief Title: Efficacy of Laser Therapy for Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Science and Technology, Yemen (Other)
Responsible Party: Principal Investigator, Amani Abdulhakeem Alsharani, Assistant Lecturer and principal investigator, University of Science and Technology, Yemen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLT-UST-YEMEN
Record Dates: First submitted 2025-05-24; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Disease
Keywords: Periodontal disease; Diode laser; Non-surgical periodontal therapy; Gingival crevicular fluid; IL-1B; IL-6; IL-8; TNF; Laser dentistry; Periodontitis; Yemen
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Curettage; Single Person

STUDY DESIGN:
Intervention Model Description: This is a three-arm parallel assignment study comparing the effects of different periodontal treatments in patients with periodontitis. Participants were randomly assigned to one of the following groups: (1) scaling and root planing (SRP) alone, (2) SRP combined with high-power diode laser, or (3) SRP combined with low-power diode laser. The study aimed to evaluate changes in clinical periodontal parameters and inflammatory cytokine levels in gingival crevicular fluid at baseline, 1 month, and 3 months after treatment.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- scaling and root planning (SRP) (Active Comparator): Patients receive only subgingival curettage by curettes and ultrasonic scaler
  Interventions: Procedure: Curettage (SRT) only
- High Diode Laser (H D Laser) (Experimental): Patients recieved high power diode laser (2W) after curettage to pocket disinfection and tissue healing
  Interventions: Procedure: High power diode laser + SRT; Procedure: Curettage (SRT) only
- Low Diode Laser (L D Laser) (Experimental): Low power laser(0. 5W) is applicated to patient after curettage
  Interventions: Procedure: Low diode diode laser + SRT; Procedure: Curettage (SRT) only

INTERVENTIONS:
Procedure: High power diode laser + SRT — 2W laser will be applied to periodontal pockets
  Arms: High Diode Laser (H D Laser)
Procedure: Low diode diode laser + SRT — A 0.5W low laser is applicated to periodontal pockets after mechanical debridement
  Arms: Low Diode Laser (L D Laser)
Procedure: Curettage (SRT) only — Mechanical debridement for pocket

SUMMARY:
The aim of this study is to evaluate the efficacy of diode laser in addition to periodontal treatment in periodontitis patients and to investigate their effects on gingival crevicular fluid (GCF) cytokine levels before and after treatment, among some Yemeni individuals in Sana'a city.

DETAILED DESCRIPTION:
This study aims to compare the clinical and immunological effects of traditional mechanical debridement alone versus combined treatment with diode laser (high and low power). The clinical parameters include Plaque Index (PI), Gingival Index (GI), Periodontal Pocket Depth (PPD), and Clinical Attachment Loss (CAL). Immunological parameters include IL-1β, IL-6, IL-8, and TNF-α levels in GCF. Participants will be selected from the Yemeni population residing in Sana'a City. The study will include a control group receiving conventional therapy and two test groups receiving diode laser therapy with high and low intensity settings, respectively. Measurements will be recorded at baseline (T0), one month after treatment (T1), and three months post-treatment (T2).

The goal is to determine whether adjunctive diode laser therapy provides additional clinical and immunological benefits compared to conventional treatment alone.

ELIGIBILITY:
Inclusion Criteria:

Only patients meeting the following criteria will be enrolled into the study:

* Patient with generalized periodontitis (BOP and PPD ≥ 4 mm).
* Age group of 25-58 years old of periodontitis patients with at least 20 teeth present.

Exclusion Criteria:

* Smoker and qat chewer patients.
* Pregnant and lactating women.
* Patients take medications which might influence the periodontal tissue state.
* Patients having systemic health disorders which affect the periodontium by history.
* Patients who received periodontal treatment or antibiotic therapy 3 months before the study.

VI. Patient wearing intra-oral appliance or with dental prosthesis. :

-

Ages: 25 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in clinical periodontal parameters (Plaque Index) | Baseline,1 month, 3months after treatment
  Clinical evaluation of plaque index will be performed at three points before treatment (T0), 1 month (T1) anD 3 months (T2) after treatment to evaluate periodontal improvement
Change in clinical periodontal parameters (Gingival Index) | Baseline,1 month, 3months after treatment
  Clinical evaluation of gingival index will be performed at three points before treatment (T0), 1 month (T1) anD 3 months (T2) after treatment to evaluate periodontal improvement
Change in clinical periodontal parameters (Periodontal Pocket Depth) | Baseline,1 month, 3months after treatment
  Clinical evaluation of periodontal pocket depth will be performed at three points before treatment (T0), 1 month (T1) anD 3 months (T2) after treatment to evaluate periodontal improvement
Change in clinical periodontal parameters (Clinical attachment level) | Baseline,1 month, 3months after treatment
  Clinical evaluation of clinical attachment level will be performed at three points before treatment (T0), 1 month (T1) anD 3 months (T2) after treatment to evaluate periodontal improvement

SECONDARY OUTCOMES:
Change in interleukin-6 (IL-6) levels in GCF | Baseline,1 month, 3months after treatment
  Levels of interleukin-6 (IL-6) in gingival crevicular fluid (GCF) will be measured at baseline, 1 month, and 3 months after treatment to assess immune response to o assess immune response to periodontal therapy.
Change in interleukin-1B (IL-1B) levels in GCF | Baseline,1 month, 3months after treatment
  Levels of interleukin-1 beta (IL-1β) in gingival crevicular fluid (GCF) will be measured at baseline, 1 month, and 3 months after treatment to assess immune response to periodontal therapy
Change in interleukin-8 (IL-8) levels in GCF | Baseline,1 month, 3months after treatment
  Levels of interleukin-8 (IL-8) in gingival crevicular fluid (GCF) will be measured at baseline, 1 month, and 3 months after treatment to assess immune response to o assess immune response to periodontal therapy.
Change in tumor necrosis factor-alpha (TNF-α) levels in GCF | Baseline,1 month, 3months after treatment
  Levels of tumor necrosis factor-alpha (TNF-α) in gingival crevicular fluid (GCF) will be measured at baseline, 1 month, and 3 months after treatment to assess immune response to o assess immune response to periodontal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Waddah N Al-Hajj, Assoc prof, Study Chair — Faculty of dentistry -Thamar university

IPD SHARING:
Plan to Share IPD: Yes
"De-identified individual participant data (IPD) including demographic information, treatment assignment, clinical outcomes, and cytokine levels will be shared. The data will be made available to qualified researchers for non-commercial academic use after publication of the primary results."
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication, available for 5 years
Access Criteria: Data will be shared upon reasonable request to the corresponding author via email
URL: https://www.ust.edu.ye

REFERENCES:
- See also: University of Science and Technology - Yemen official site — https://www.ust.edu.ye
- Available data/document: Study Protocol — http://www.ust.edu.ye — De-identified data including patient demographics, treatment allocation (scaling only, scaling + high-power diode laser, scaling + low-power diode laser), changes in periodontal pocket depth, and levels of cytokines (IL-1β, IL-6, IL-8, TNF-α) will be made available. Data access will be granted upon reasonable request submitted to the corresponding author via email at: aamanialsharani.aa@gmail.com.